CLINICAL TRIAL: NCT01870011
Title: A Comparison of Propofol Based Total Intravenous Anesthesia and Desflurane Based Balanced Anesthesia on Renal Protection During Deceased Brain Dead Donor Kidney Transplantation - A Prospective, Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2013-0208
Record Dates: First submitted 2013-05-30; First posted 2013-06-05 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Disease
Keywords: Propofol, renal protection, kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desflurane balanced anesthesia group (Experimental)
  Interventions: Drug: Desflurane balanced anesthesia
- Propofol total intravenous anesthesia group (Active Comparator)
  Interventions: Drug: Propofol total intravenous anesthesia

INTERVENTIONS:
Drug: Desflurane balanced anesthesia — Desflurane balanced anesthesia induced with thiopental sodium, remifentanil and atracurium and maintained with remifentanil target controlled infusion and desflurane inhalation
  Arms: Desflurane balanced anesthesia group
Drug: Propofol total intravenous anesthesia — Propofol total intravenous anesthesia induced with propofol, remifentanil and atracurium and maintained with remifentanil and propofol target controlled infusion
  Arms: Propofol total intravenous anesthesia group

SUMMARY:
Renal ischemia/reperfusion (I/R)-induced injury is known to be associated with immediate and long-term kidney dysfunction after renal transplantation. Protecting the kidney against I/R injury and maintaining renal function during renal transplant surgery is therefore very important in order to improve post-operative outcome. This purpose of this study is to investigate whether propofol anesthesia done in both kidney donors and recipients during deceased brain dead donor kidney transplantation is effective in reducing renal I/R injury via its antioxidant and antiinflammatory properties and improve post-transplant outcome compared to desflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult deceased brain dead kidney donors and recipients scheduled for renal transplantation

Exclusion Criteria:

1. Donor exclusion criteria:

(1) Refusal of legal guardian

2. Recipient exclusion criteria:

1. Patient refusal
2. Hypersensitivity to propofol, soybeans or peanuts
3. History of vitamin C or E intake within 5 days before surgery
4. History of acute myocardial infarct within 6 months before surgery
5. Congestive heart failure (NYHA III-IV)
6. Autoimmune disease patients
7. BMI over 30 kg/m2
8. Left ventricular ejection fraction less than 35% upon preoperative echocardiography

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The difference in inflammatory markers of recipients between groups during and after renal transplantation (CRP, WBC differential count, IL-6, TGF-β) | Inflammatory markers are evelauted immediately after anesthesia induction, right before kidney extraction and 1 hour after kidney extraction
  1. Kidney donor: Inflammatory markers are evaluated immediately after anesthesia induction, right before kidney extraction and 1 hour after kidney extraction
  2. Kidney recipient:
  (1) Inflammatory markers: Immediately after anesthesia induction, 2 and 24 hours after reperfusion (2) Renal function markers: Before anesthesia, 2 hours after reperfusion, immediate post-op, 24 and 48 hours postoperatively

SECONDARY OUTCOMES:
The difference in renal function of kidney recipients between groups after renal transplantation (BUN/Cr, cystatin C, NGAL) | immediately after anesthesia induction, right before kidney extraction and 1 hour after kidney extraction
  1. Kidney donor: Inflammatory markers are evaluated immediately after anesthesia induction, right before kidney extraction and 1 hour after kidney extraction
  2. Kidney recipient:
  (1) Inflammatory markers: Immediately after anesthesia induction, 2 and 24 hours after reperfusion (2) Renal function markers: Before anesthesia, 2 hours after reperfusion, immediate post-op, 24 and 48 hours postoperatively

OTHER OUTCOMES:
The difference in global oxidative stress markers of recipients between groups during and after renal transplantation (Free Oxygen Radicals Testing, Free Oxygen Radial Defense) | changes of Global oxidative stress markers from Immediately after anesthesia induction to 2 hours after reperfusion
  1. Kidney donor: Inflammatory markers are evaluated immediately after anesthesia induction, right before kidney extraction and 1 hour after kidney extraction
  2. Kidney recipient:
  (1) Inflammatory markers: Immediately after anesthesia induction, 2 and 24 hours after reperfusion (2) Renal function markers: Before anesthesia, 2 hours after reperfusion, immediate post-op, 24 and 48 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea